CLINICAL TRIAL: NCT01735643
Title: Spielend zu Mehr Bewegung - Lebensstilintervention Durch Das Interaktive Video-spiel "Wii Fit Plus" Bei Personen Mit Typ-2-Diabetes Mellitus
Brief Title: Lifestyle Intervention With an Interactive Video Game for Type 2 Diabetes Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Nintendo of Europe GmbH (Unknown)
Responsible Party: Principal Investigator, Stephan Martin, MD, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wii study
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; physical activity; lifestyle change; motivation; patient empowerment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interactive videogame intervention (Experimental)
  Interventions: Device: interactive videogame Wii Fit Plus
- waiting group (Experimental)
  Interventions: Other: waiting

INTERVENTIONS:
Device: interactive videogame Wii Fit Plus — Use of the interactive videogame Wii Fit Plus für 12 weeks.
  Other Names: Wii Fit Plus
  Arms: interactive videogame intervention
Other: waiting — waiting for 12 weeks
  Arms: waiting group

SUMMARY:
Due to overweight and unhealthy lifestyle the number of patients with type 2 diabetes mellitus is increasing. Although in early phases the disease might be successfully treated by lifestyle change patients lack for motivation. Instead of increasing anti-diabetic medication a highly motivational system with low inhibition threshold is needed. Therefore, the investigators analyzed if regular use of the interactive videogame Wii Fit Plus over 12 weeks is able to improve HbA1c and weight in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Patients with type 2 diabetes were recruited via treating physicians or articles in magazines and newspapers. Participants were randomized in an intervention and a control group. The intervention group was sent the Wii, the balance board and the interactive video game Wii Fit Plus and were instructed to use these items 30 minutes each day during the next 12 weeks. The control group got the items 12 weeks later. At begin and after 12 weeks of intervention participants (and additionally for the control group: after 12 weeks of waiting phase) sent their health parameters, which had been measured in the context of the disease management program type 2 diabetes as well as questionnaires about physical activity and quality of life to the study center.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* diabetes duration < 5 years
* age 50-75 years
* body mass index > or equal to 27 kg/m2
* participating in the disease management programme type 2 diabetes mellitus
* physical and mental able for study participation

Exclusion Criteria:

* insulin or antidiabetic medication (exception: Metformin and DPP-IV-Inhibitors)
* regular physical activity
* depression
* tumors
* change of smoking status during the past 6 months or during the study
* participation in other studies during the past 6 months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2011-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks

SECONDARY OUTCOMES:
weight | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, MD, Principal Investigator — West German Center of Diabetes and Health
Locations (1):
- West German Center of Diabetes and Health, Düsseldorf, Germany

REFERENCES:
- [Derived] Kempf K, Martin S. Autonomous exercise game use improves metabolic control and quality of life in type 2 diabetes patients - a randomized controlled trial. BMC Endocr Disord. 2013 Dec 10;13:57. doi: 10.1186/1472-6823-13-57. PMID 24321337
- See also: Affiliation homepage — http://www.vkkd-kliniken.de